CLINICAL TRIAL: NCT00631137
Title: A Randomized, Controlled Comparative Trial to Determine if Testosterone Gel Prevents Steroid Related Weakness in Brain Cancer Patients
Brief Title: Testosterone Gel in Preventing Weakness Caused by Steroid Therapy in Men With Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to low accrual.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: J0634; P30CA006973 (NIH); JHOC-J0634 (Other: Johns Hopkins University SKCCC); NA_00003125 (Other: Johns Hopkins University IRB); CDR0000584274 (Other: other)
Record Dates: First submitted 2008-03-06; First posted 2008-03-07 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Brain and Central Nervous System Tumors; Musculoskeletal Complications
Keywords: musculoskeletal complications; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Arm 1: Control Group (Placebo Comparator): whey protein powder
  Interventions: Dietary Supplement: whey powder protein
- ARM 2 : Treatment Group (Active Comparator): Testosterone Gel (10g pouch/day) applied to skin
  Interventions: Drug: testosterone gel applied to skin

INTERVENTIONS:
Drug: testosterone gel applied to skin — Application of testosterone gel
  Arms: ARM 2 : Treatment Group
Dietary Supplement: whey powder protein
  Arms: Arm 1: Control Group

SUMMARY:
RATIONALE: Testosterone gel may be effective in preventing or lessening muscle weakness caused by steroid therapy in men receiving glucocorticoids for newly diagnosed high-grade glioma.

PURPOSE: This randomized clinical trial is studying how well testosterone gel works in preventing weakness caused by steroid therapy in men receiving glucocorticoids for newly diagnosed high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if daily administration of testosterone gel can prevent the development or reduce the severity of muscle weakness in men receiving glucocorticoids for newly diagnosed high-grade glioma.

Secondary

* To compare the difference in percent change from baseline timed functional tests (TFT) between patients who are treated with testosterone gel and those who are not.
* To compare the difference in percent change from baseline activities of daily living as assessed by the Health Assessment Questionnaire-Disability Index (HAQ-DI) between patients who are treated with testosterone gel and those who are not.
* To compare the difference in percent change from baseline leg muscle mass as assessed by CT scan imaging between patients who are treated with testosterone gel and those who are not.
* To estimate the side effects of testosterone gel in these patients.

OUTLINE: Patients are stratified according to daily glucocorticoid dose (< 16 mg/day vs ≥ 16 mg/day), Karnofsky performance status (≤ 80% vs > 80%), and age (≤ 50 years of age vs > 50 years of age). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive oral whey protein powder once daily for 7 months.
* Arm II (treatment): Patients apply topical testosterone gel to the shoulder, upper chest, or forearm once daily for 7 months.

Patients undergo strength testing and functional testing (TFT) and complete an activities of daily living questionnaire at baseline and at 1, 3, 5, and 7 months. Patients also undergo CT scan of the leg and laboratory testing at baseline and at 3 and 7 months. Testosterone levels are obtained at baseline and at 1, 3, and 7 months.

Patients complete a daily log of their glucocorticoid dose and to affirm compliance with therapy. Major clinical events related to underlying tumor (i.e., surgery, radiotherapy, initiating chemotherapy, concurrent antiepileptic therapy, deep vein thrombosis, pulmonary embolism, transfusions, seizures, pneumonia, and other forms of infection) are also recorded.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed high-grade glioma, including the following subtypes:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Requires dexamethasone at a dose of > 4 mg/day to control symptoms of tumor-related edema at time of study enrollment AND has been on a stable dose of steroids for ≥ 5 days prior to study enrollment
* Completed ≥ 80% of prescribed radiotherapy
* Hypogonadal, defined as serum testosterone level < 350 ng/dL
* No history of prostate or breast cancer
* No benign prostatic hypertrophy requiring therapy OR AUA score of ≥ 8

  * PSA ≤ 4 ng/mL

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Able to keep daily records or has a care provider that agrees to keep daily records of drug administration
* No clinical history of congestive heart failure requiring therapy
* No psychotic disorder requiring active treatment
* No structured exercise program involving exercise for > 3 hours/week
* No polycythemia (i.e., hematocrit > 52%)

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior androgen therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaishri O. Blakeley, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: outpatient clinic
Groups:
- ARM 2 : Treatment Group: Androgel (10g pouch/day)
  testosterone gel :
  questionnaire administration :
- Arm 1: Control Group: whey protein powder
  questionnaire administration :
Period: Overall Study
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were assigned to the Control Group Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: years] | 29 |  | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Event, Defined as ≥ 50% Loss of Strength in the Hip Flexors as Assessed by Dynamometry Peak Force Measures at Baseline and at 1, 3, 5, and 7 Months
Time Frame: baseline and at 1, 3, 5, and 7 months
Population: Only 1 subject accrued. Not enough data to analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Muscle Strength Testing in Other Proximal Muscles (i.e., Knee Extensors, Knee Flexors, Arm Abductors, Elbow Extensors and Flexors, and Neck Flexors) as Assessed by Dynamometry at Baseline and at 1, 3, 5, and 7 Months
Time Frame: baseline and at 1, 3, 5, and 7 months
Population: Only 1 subject accrued. Not enough data to analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Performance on Timed Functional Tests (TFT) as Assessed at Baseline and at 1, 3, 5, and 7 Months
Time Frame: baseline and at 1, 3, 5, and 7 months
Population: Only 1 subject accrued. Not enough data to analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Leg Muscle Mass as Assessed by CT Scan at Baseline and at 3 and 7 Months
Time Frame: baseline and at 3 and 7 months
Population: Only 1 subject accrued. Not enough data to analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Activities of Daily Living as Assessed by the Health Assessment Questionnaire-Disability Index at Baseline and at 1, 3, 5, and 7 Months
Time Frame: baseline and at 1, 3, 5, and 7 months
Population: only 1 subject enrolled. Not enough to do analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Side Effects of Testosterone Gel as Assessed by Frequency of Adverse Events, Including Laboratory Abnormalities
Time Frame: while receiving treatment
Population: only 1 subject enrolled. Not enough to do analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serum Total Testosterone Levels as Assessed at Baseline and at 1, 3, and 7 Months
Time Frame: baseline and at 1, 3, and 7
Population: only 1 subject enrolled. Not enough to do analysis
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: through study completion, up to 1 year
Description: The definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definition.
Arm/Group | ARM 2 : Treatment Group | Arm 1: Control Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 2 : Treatment Group (N=1) | Arm 1: Control Group (N=0)
rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — grade 1

LIMITATIONS AND CAVEATS:
early termination, leading to only 1 subject enrolled, hence could NOT do data analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes